CLINICAL TRIAL: NCT06755281
Title: Risk-stratified Testing for Safe Removal of Penicillin Allergy Labels
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Deniz Göcebe (Other)
Responsible Party: Sponsor-Investigator, Deniz Göcebe, Dr. med. Deniz Göcebe, University Hospital Heidelberg
Organization: University Hospital Heidelberg (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: S-656/2024
Record Dates: First submitted 2024-12-22; First posted 2025-01-01 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Penicillin Allergy; Hypersensitivity, Immediate; Hypersensitivity, Delayed; Hypersensitivity Response
Keywords: PEN-FAST; penicillin allergy; allergy delabeling
MeSH Terms: conditions — Hypersensitivity, Immediate; Hypersensitivity, Delayed | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Direct drug provocation test (Experimental)
  Interventions: Other: Direct Oral challenge
- Standard of care (Active Comparator): Standard of care Skin testing and measurement of allergen-specific IgE, if negative, drug provocation test.
  Interventions: Other: standard of care

INTERVENTIONS:
Other: Direct Oral challenge — Patients will receive a 1-step or 2-step challenge with the suspected penicillin and will be monitored for any allergic reaction within the first four hours. Patients will be instructed to contact the hospital after the drug provocation test to inquire delayed allergic reactions.
  Arms: Direct drug provocation test
Other: standard of care — The patient will receive skin prick test and patch test (if a delayed allergy is suspected). Allergen-specific IgE will be measured. If all negative, drug provocation tets will be performed identical to the experimental group.
  Arms: Standard of care

SUMMARY:
The aim of this clinical trial is to analyze the negative predictive capacity and safety of risk-stratified direct drug provocation tests for patients with self-reported penicillin allergies. Patients reporting immediate or delayed penicillin allergies and defined as low-risk by the PEN-FAST score will receive drug provocation tests without prior skin testing.

DETAILED DESCRIPTION:
The PEN-FAST clinical decision rule is an internationally validated scoring system (0-5 points) that identifies low-risk patients (= a score of 0-2 points) with self-reported penicillin allergies with a negative predictive value (NPV) of over 95%. Performing direct drug provocation tests without prior skin testing on these low-risk patients was shown to be non-inferior in terms of safety and prediction of immediate allergic reactions. However, several studies have questioned the negative predictive capacity of the PEN-FAST score. In these studies, misclassifications of the PEN-FAST score were mainly based on positive skin test findings that can show false-positive results.

This study aims to validate the NPV and safety of direct drug provocation tests using the PEN-FAST score.

Participants with a PEN-FAST score of 0-2 points will directly receive a two-dose challenge (50%-50%) or single challenge (100%) with the culprit penicillin and will be monitored for at least 4 hours. No skin tests will be performed prior to the drug provocation test. Patients will be instructed to contact the hospital after the drug provocation test to monitor any delayed allergic reactions.

The outcomes will be compared to those of patients with a PEN-FAST score of 0-2 points who do not wish to skip the skin tests and who will, in parallel, receive the standard-of-care testing.

Currently, this study is approved as a single-site study.

ELIGIBILITY:
Inclusion Criteria:

1. Adult outpatients or inpatients with a penicillin allergy label
2. Willing and able to give consent.
3. PEN-FAST score of 0-2 points

Exclusion Criteria:

1. Age <18 years
2. Concurrent immunosuppressive therapy with 20 mg of prednisolone per day or steroid equivalent
3. Concurrent antihistamine therapy
4. Pregnancy
5. Significantly impaired general condition
6. Unstable or therapeutically inadequately controlled bronchial asthma
7. History of stem cell transplantation
8. History of acute interstitial nephritis
9. Chronic urticaria
10. Mastocytosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
The difference in the proportion of patients with any positive finding in skin tests, allergen-specific IgE or drug provocation test between the two groups | 7 days
  Percentage of subjects that retain their allergy label as they show at least one positive finding in skin tests, allergen-specific IgE or drug provocation test.

SECONDARY OUTCOMES:
Negative predictive capacity of skin tests and allergen-specific IgE | 7 days
  Negative predictive values of each test alone and combined
Analysis of medical and allergic history | 1 day
  (supposed) allergic symptoms
Penicillin allergy label | 1 day
  Identification of culprit penicillin
Analysis of demographic data | 1 day
  Age, sex
Analysis of adverse reactions | 7 days
  Detailed analysis of any (supposed) allergic reactions following drug provocation test
Analysis of medical and allergic history | One day
  year of (supposed) allergic reaction
Analysis of medical and allergic history | One day
  time between administration and (supposed) allergic reaction
Analysis of medical and allergic history | One day
  treatment required for (supposed) allergic reaction
Analysis of medical and allergic history | One day
  current medication
Analysis of internal hospital risk stratification system | One day
  Measurement of score of internal hospital risk stratification system
Analysis of medical and allergic history | One day
  (supposed) allergic symptoms

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University Hospital Heidelberg, Dermatology, Heidelberg, Baden-Wurttemberg
  - University Hospital Heidelberg, Division of Infectious Diseases and Tropical Medicine, Heidelberg, Baden-Wurttemberg

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article that is planned to be published, after deidentification.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who offer a well-structured and scientifically sound approach to realizing the objectives detailed in the approved proposal.

REFERENCES:
- [Background] Copaescu AM, Vogrin S, James F, Chua KYL, Rose MT, De Luca J, Waldron J, Awad A, Godsell J, Mitri E, Lambros B, Douglas A, Youcef Khoudja R, Isabwe GAC, Genest G, Fein M, Radojicic C, Collier A, Lugar P, Stone C, Ben-Shoshan M, Turner NA, Holmes NE, Phillips EJ, Trubiano JA. Efficacy of a Clinical Decision Rule to Enable Direct Oral Challenge in Patients With Low-Risk Penicillin Allergy: The PALACE Randomized Clinical Trial. JAMA Intern Med. 2023 Sep 1;183(9):944-952. doi: 10.1001/jamainternmed.2023.2986. PMID 37459086
- [Background] Trubiano JA, Vogrin S, Chua KYL, Bourke J, Yun J, Douglas A, Stone CA, Yu R, Groenendijk L, Holmes NE, Phillips EJ. Development and Validation of a Penicillin Allergy Clinical Decision Rule. JAMA Intern Med. 2020 May 1;180(5):745-752. doi: 10.1001/jamainternmed.2020.0403. PMID 32176248